CLINICAL TRIAL: NCT04606225
Title: The Role of the Renin-angiotensin System in Emotion-memory Interactions
Brief Title: Losartan Effects on Emotion-memory Interaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-74
Record Dates: First submitted 2020-10-09; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: Losartan; Emotion-memory interaction
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Drug: Losartan
  Interventions: Drug: Losartan
- Placebo group (Placebo Comparator): Drug: Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Losartan — administration of losartan (50 mg) (oral) Cozaar Oral Tablet
  Other Names: Cozaar Oral Tablet
  Arms: Losartan group
Drug: Placebo Oral Tablet — administration of placebo (oral)
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate whether a single dose of losartan (50 mg) can affect emotion-memory interaction in healthy humans and its underlying neural mechanisms.

DETAILED DESCRIPTION:
Animal models and initial findings in humans suggest a role of the renin-angiotensin system in cognitive and emotional processes. Accumulating evidence demonstrates modulatory effects of the angiotensin antagonist losartan in the domains of memory and emotional processing. Against this background the present study aims to investigate the behavioral and neural effects of a single dose of losartan on emotional processing and emotion-memory integration in healthy subjects. In a double-blind, between-subject, placebo-controlled pharmaco-fMRI experiment, 60 male participants will be randomized to a single dose of losartan (50 mg) or placebo, and encode emotional pictures during fMRI (scheduled 90 minutes after drug administration). Then 24 hours post fMRI participants will finish a surprise recognition memory test to estimate the emotion effects on subsequent memory.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness
* Normal or corrected-normal version

Exclusion Criteria:

* History of head injury
* Medical or psychiatric illness
* Hypertension
* General cardio-vascular alteration or diseases
* Allergy against medications
* Visual or motor impairments
* Claustrophobia
* Drug addiction
* Nicotine dependence
* FMRI contradictions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
fMRI-based indices of neural activity during processing of emotional stimuli will be compared between the treatment groups | 120 to 150 minutes after treatment
  Neural activation during processing of emotional pictures will be assessed by functional magnetic resonance imaging (fMRI). The fMRI data will be analyzed by a Generalized Linear Model approach. Effects of treatment will be determined by comparing the losartan-treated group with the placebo-treated group.
fMRI-based indices of neural activity for subsequently successfully remembered as compared to non-remembered stimuli will be compared between the treatment groups | 120 to 150 minutes after treatment
  Neural activation for stimuli that are successfully remembered after an interval of 24hours will be compared to stimuli that are not successfully remembered. Neural activity between the subsequently remembered and non-remembered stimuli will be assessed by functional magnetic resonance imaging (fMRI) acquired during the initial encoding of the stimuli. The fMRI data will be analyzed by a Generalized Linear Model approach. Effects of treatment will be determined by comparing the losartan-treated group with the placebo-treated group.

SECONDARY OUTCOMES:
Self-Assessment Manikin (SAM) ratings of arousal of the stimuli will be compared between the treatment groups | 120 to 150 minutes after treatment
  During the fMRI participants will rate the emotional arousal of each presented picture by means of the Self-Assessment Manikin (SAM). The assessment ranges from 1-5, with 1 referring to very low arousal while 5 refers to a very high arousal. The effects of treatment on arousal will be examined by comparing the losartan-treated with the placebo-treated group by means of a Generalized Linear Model approach.
Self-Assessment Manikin (SAM) ratings of valence of the stimuli will be compared between the treatment groups | 120 to 150 minutes after treatment
  During the fMRI participants will rate the emotional valence of each presented picture by means of the Self-Assessment Manikin (SAM). The assessment ranges from 1-5, with 1 referring to very negative valence, while 5 refers to a very positive valence. The effects of treatment on valence will be examined by comparing the losartan-treated with the placebo-treated group by means of a Generalized Linear Model approach.
Memory performance in terms of correctly recognized stimuli will be compared between the treatment groups | 24 hours after treatment
  24 hours after the fMRI assessment subjects will be re-exposed to the stimuli that were presented during the fMRI and new stimuli. Subjects have to indicate for each stimulus whether it has been shown during fMRI. Memory performance in terms of correct responses will be computed and compared between the losartan-treated with the placebo-treated group by means of a Generalized Linear Model approach.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu T, Zhou X, Jiao G, Zeng Y, Zhao W, Li J, Yu F, Zhou F, Yao S, Becker B. Angiotensin Antagonist Inhibits Preferential Negative Memory Encoding via Decreasing Hippocampus Activation and Its Coupling With the Amygdala. Biol Psychiatry Cogn Neurosci Neuroimaging. 2022 Oct;7(10):970-978. doi: 10.1016/j.bpsc.2022.05.007. Epub 2022 May 30. PMID 35654318